CLINICAL TRIAL: NCT06177821
Title: Feasibility of Water Vaporization (Rezum®) for Patients With ≥ 30 and < 80 ml With Moderate-severe LUTS to Establish the Surgical Principles for Prominent or Non-prominent Median Lobe Enlargement: A Single-center, Prospective, Pilot Study
Brief Title: Rezum for 30-80ml Patients With Moderate-severe LUTS to Study Surgical Principles for Median Lobe Enlargement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Cho, M.D., Ph.D., Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REZUM
Record Dates: First submitted 2023-11-30; First posted 2023-12-20 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Prostatic Hyperplasia of the Medial Lobe
Keywords: median lobe enlargement; lower urinary tract symptoms; International Prostate Symptoms Score
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, 5 seconds (Experimental): Patients with benign prostatic hyperplasia featuring a small median lobe enlargement will be allocated to the 5-second Rezum therapy group.
  Interventions: Device: Rezum®
- Group B, 9 seconds (Experimental): Patients with benign prostatic hyperplasia featuring a big prominent median lobe enlargement will be allocated to the 9-second Rezum therapy group.
  Interventions: Device: Rezum®

INTERVENTIONS:
Device: Rezum® — Rezum® Water vaporization device

SUMMARY:
This study was created to determine the safety and efficacy of treating prostatic hyperplasia with or without prominent median lobe enlargement with the REZUM technique. The systematic implementation of decisions for the location, vapor time, and the number of injections contributes to the Rezum procedure configuration for the median lobe treatment being safer and standardizer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 85 years who have been diagnosed with benign prostatic hyperplasia at Seoul National University Hospital and are scheduled to undergo endoscopic surgery.
* benign prostatic hyperplasia ≥ 30 and < 80 ml
* Patients who have given written informed consent to participate in the study according to their age
* A urinary symptom score (International ProstateSymptom Score [IPSS] moderated (8-19 points) to severe (20-35 points)
* Measured Postvoiding Residual (PVR) <250 mL

Exclusion Criteria:

* History of prostate or bladder cancer, neurogenic bladder, bladder calculus, or clinically significant bladder diverticulum
* Active infection, treatment for chronic prostatitis
* Diagnosis of urethral stricture, meatal stenosis or bladder neck contracture, damaged external urinary sphincter, stress urinary incontinence, post-void residual >300 mL or urinary retention, or prior prostate surgery
* Men taking anticoagulants or on bladder anticholinergics or with severe cardiovascular disease
* PSA greater than 4.0 ng/ml (unless prostate cancer was ruled out by biopsy)
* Allergy to device materials, immune suppressants or corticosteroids use, and serious medical or mental illness.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2024-06-17 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
age | prior to procedure
  patient's records
Gender | prior to procedure
  patient's records
height | prior to procedure
  meters
weight | prior to procedure
  kilograms
Medical history | prior to procedure
  patient's records
Surgical history | prior to procedure
  patient's records
Date of consent | prior to procedure
  patient's records
Eastern Cooperative Oncology Group | prior to procedure
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
complications | prior to procedure
  patient's records
medications used at the time of pre-consent | prior to procedure
  patient's records
drug allergies | prior to procedure
  patient's records
prostate specific antigen | prior to procedure, 3 month after surgery
  patient's records, ng/ml
Protein | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, mg/dl
pH | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis
occult blood | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, Negative or positive
white blood cell : Urinalysis | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, Quantity
glucose | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, mg/dl
red blood cell | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, Quantity
Bacteria | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Urinalysis, Quantity
Sodium | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mEq/L
Chloride | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mEq/L
calcium | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dL
Phosphorus | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dL
uric acid | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dl
blood urea nitrogen | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dl
creatinine | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dL
C-reactive protein | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, mg/dl
White blood cell : Blood tests | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, quantity
Hemoglobin | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, g/dl
Platelet | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, 10^3/μL
Prostate specific antigen | prior to procedure, 1-2 weeks after injection, 3 month after surgery
  Blood tests, ng/ml
Prostate Ultrasound | prior to procedure, 3 month after surgery
  patient's records
Uroflowmetry | prior to procedure, 3 month after surgery
  patient's records, ml/sec
International Prostate Symptom Score | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  0 to 7 points: Mild symptoms 8 to 19 points: Moderate symptoms 20 to 35 points: Severe symptoms
Incontinence Severity Index | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  Slight (1-2) Moderate (3-6) Severe (8-9) Very severe (12)
Overactive Bladder Symptom Score | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  1. How many times do you typically urinate from waking in the morning until sleeping at night?
  7 or less 8 to 14 15 or more 2. How many times do you typically wake up to urinate from sleeping at night until waking in the morning?
  0
  1 2 3 or more 3. How often do you have a sudden desire to urinate, which is difficult to defer?
  Not at All less than once a week once a week or more about once a day 2 to 4 times per day 5 times a day or more 4. How often do you leak urine, because you cannot defer the sudden desire to urinate?
  Not at All less than once a week once a week or more about once a day 2 to 4 times per day 5 times a day or more
Male Sexual Health for assessing ejaculatory dysfunction | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  1. In the last month, without using drugs like Viagra, how often have you been able to get an erection when you wanted to? 5 All of the time 4 Most of the time 3 About half of the time 2 Less than half of the time 1 None of the time 0 Used Viagra or similar drug with every sexual encounter
  2. In the last month, if you were able to get an erection without using drugs like Viagra, how often were you able to stay hard as long as you wanted to? 5 All of the time 4 Most of the time 3 About half of the time 2 Less than half of the time 1 None of the time 0 Used Viagra or similar drug with every sexual encounter
  3. In the last month, if you were able to get an erection, without using drugs like Viagra, how would you rate the hardness of your erection? 5 Completely hard 4 Almost completely hard 3 Mostly hard, but can be slightly bent 2 A little hard, but bends easily 1 Not at all hard 0 Used Viagra or similar drug with every sexual encounter
International Index of Erectile Function | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  The IIEF-5 Questionnaire (SHIM)Score for Erectile Dysfunction1-7: Severe8-11: Moderate12-16: Mild-moderate17-21: Mild22-25: No Erectile Dysfunction Survey.
McGill Pain Questionnaire | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  The interpretation of the questionnaire is pretty basic: the higher the score, the higher the pain level. The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain.
Brief Pain Inventory | prior to procedure, admission, 1-2 weeks after injection, 3 month after surgery
  Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Treatment Satisfaction-Visual Analogue Scale | 1-2 weeks after injection, 3 month after surgery
  0. No, not at all satisfied. 10. Yes, completely satisfied.
Patient Global Impression of Improvement | 1-2 weeks after injection, 3 month after surgery
  Very much better 1 Much better 2 A little better 3 No change 4 A little worse 5 Much worse 6 Very much worse 7
transrectal sonography of the prostate | prior to procedure, 3 month after surgery
  Ultrasound examination
transrectal ultrasound | prior to procedure
  Ultrasound examination
Postvoiding Residual | prior to procedure, 3 month after surgery
  uroflowmetry
Post-surgery complications | 1-2 weeks after injection, 3 month after surgery
  patient's records

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The datasets used during the current study are available from the corresponding author on request.